CLINICAL TRIAL: NCT00362609
Title: A Multicenter, Open-Label, PK, PD and Safety Study of Pantoprazole Delayed-Release Granules Administered as a Suspension in Neonates and Preterm Infants With a Clinical Diagnosis of GERD
Brief Title: Study Evaluating Pantoprazole in Neonates and Preterm Infants With GERD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3001B3-331, 3001B3-335
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Results first posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-04

CONDITIONS: Gastroesophageal Reflux
Keywords: Safety
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

ARMS (2):
- Low dose (Active Comparator)
  Interventions: Drug: pantoprazole
- High dose (Active Comparator)
  Interventions: Drug: pantoprazole

INTERVENTIONS:
Drug: pantoprazole

SUMMARY:
The purpose of this study is to determine whether or not consistent drug levels can be achieved in infants with presumed Gastroesophageal Reflux Disease.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients
* Presumed diagnosis of GERD
* Term or post-term infants within the neonatal period less than 28 days or preterm infants with a corrected gestational age of less than 44 weeks

Exclusion Criteria:

* cardiovascular instability
* clinically significant laboratory abnormalities
* use of warfarin, carbamazepine, phenytoin, or rifampin

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2006-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For South Africa, ZAFinfo@wyeth.com; Trial Manager, Principal Investigator — For Australia, medinfo@wyeth.com; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com; Trial Manager, Principal Investigator — For Italy, descresg@wyeth.com; Trial Manager, Principal Investigator — For Switzerland, med@wyeth.com
Locations (70):
- United States (45):
  - Phoenix, Arizona
  - Loma Linda, California
  - Oakland, California
  - Orange, California
  - Sacramento, California
  - San Diego, California
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Miami, Florida
  - Sunrise, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Lexington, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Flint, Michigan
  - Omaha, Nebraska
  - Camden, New Jersey
  - New Brunswick, New Jersey
  - Newark, New Jersey
  - Albany, New York
  - Brooklyn, New York
  - New York, New York
  - The Bronx, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Danville, Pennsylvania
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Richmond, Virginia
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Brisbane, Australia
- Belgium (2):
  - Edegem
  - Leuven
- Canada (5):
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
- Paris, France
- Germany (3):
  - Bochum
  - Osnabrück
  - Potsdam
- Italy (3):
  - Brescia
  - Napoli
  - Roma
- Rotterdam, Netherlands
- Poland (3):
  - Bydgoszcz
  - Krakow
  - Lublin
- South Africa (5):
  - Panorama, CPT
  - Pietermaritzburg, KwaZulu-Natal
  - Durban
  - Overport
  - Pretoria
- Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in multiple countries worldwide from July 2006 to December 2007.
Pre-assignment Details: Patients were screened for up to 5 days.
Groups:
- 1.25 mg Pantoprazole: 1.25 mg of pantoprazole granules daily for at least 5 days. This dosing corresponds to approximately 0.6 mg/kg
- 2.5 mg Pantoprazole: 2.5 mg of pantoprazole granules daily for at least 5 days. This dose corresponds to approximately 1.2 mg/kg
Period: Overall Study
Arm/Group | 1.25 mg Pantoprazole | 2.5 mg Pantoprazole
Started | 19 | 40
Completed | 19 | 38
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.25 mg Pantoprazole | 2.5 mg Pantoprazole | Total
Number analyzed (Participants) | 19 | 40 | 59
Age Continuous [Mean (Standard Deviation); unit: weeks (postnatal age)] | 8.63 (4.86) | 7.70 (4.20) | 8.00 (4.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 18
  Male | 14 | 27 | 41

OUTCOME MEASURES:

1. Primary Outcome: Variance of Oral Bioavailability
Description: Samples were divided between 2 groups for each dose: Group A at baseline, 2, 8, 18 hours; Group B at baseline, 1, 4, 12 hours to reduce the number of blood draws per infant. The variance of oral bioavailability was assessed to determine if further PK assessment was appropriate. It would be considered highly variable if the square root of the sum of the standard deviation squares of the area under the concentration-time curves from time zero to the time of the last quantifiable concentration (AUCT) for group A and Group B divided by the sum of the mean AUCT for group A and Group B was >1.2.
Time Frame: 1 day
Population: Single dose PK Valid-For Efficacy patients (defined as those without any major protocol violations who completed the single-dose PK determinations and taken the test article on the date the PK samples were taken). 2 poor metabolizers were excluded from this analysis.
Measure: Number; unit: ratio
Arm/Group | 1.25 mg Pantoprazole | 2.5 mg Pantoprazole
Number analyzed (Participants) | 19 | 21
ratio | 1.07 (2.59) | 0.74 (2.29)

2. Secondary Outcome: Area Under the Concentration-time Curve (AUC)
Description: AUC is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption. AUC was estimated from population pharmacokinetic (PK) modeling.
Time Frame: Baseline to 24 hours post dose on Day 1
Population: Single dose PK Valid-For-Efficacy patients (defined as those without any major protocol violations who completed the single-dose PK determinations and took the test article on the date the PK samples were taken) who also had measurable concentrations over the period of observation. 2 poor metabolizers were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | 1.25 mg Pantoprazole | 2.5 mg Pantoprazole
Number analyzed (Participants) | 14 | 19
ng*hr/mL | 3540 (2820) | 7270 (5304)

3. Secondary Outcome: Apparent Oral Clearance (Cl/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling.
Time Frame: 1 day
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/hr/kg
Arm/Group | 1.25 mg Pantoprazole | 2.5 mg Pantoprazole
Number analyzed (Participants) | 14 | 19
L/hr/kg | 0.21 (0.12) | 0.23 (0.21)

4. Secondary Outcome: Half Life
Description: Half life is the time required for half the quantity of absorbed drug to be metabolized or eliminated by normal biological processes. Half life was estimated from population pharmacokinetic (PK) modeling.
Time Frame: 1 day
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1.25 mg Pantoprazole | 2.5 mg Pantoprazole
Number analyzed (Participants) | 14 | 19
hours | 3.1 (1.5) | 2.7 (1.1)

ADVERSE EVENTS:
Arm/Group | 1.25 mg Pantoprazole | 2.5 mg Pantoprazole
Serious Adverse Events (participants affected / at risk) | 0 | 2
Other Adverse Events (participants affected / at risk) | 5 | 18
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | 1.25 mg Pantoprazole | 2.5 mg Pantoprazole
Urinary Tract Infection (Renal and urinary disorders) | 0/19 | 1/40
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0/19 | 1/40
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | 1.25 mg Pantoprazole | 2.5 mg Pantoprazole
Fever (General disorders) | 0/19 | 1/40
Hernia (General disorders) | 0/19 | 1/40
Bradycardia (Cardiac disorders) | 1/19 | 1/40
Cardiovascular physical finding (Cardiac disorders) | 1/19 | 0/40
Tachycardia (Cardiac disorders) | 0/19 | 2/40
Ventricular extrasystoles (Cardiac disorders) | 1/19 | 0/40
Constipation (Gastrointestinal disorders) | 1/19 | 2/40
Flatulence (Gastrointestinal disorders) | 0/19 | 1/40
Liver function tests abnormal (Gastrointestinal disorders) | 0/19 | 1/40
Anemia (Blood and lymphatic system disorders) | 0/19 | 5/40
Iron deficiency anemia (Blood and lymphatic system disorders) | 0/19 | 1/40
Peripheral edema (Metabolism and nutrition disorders) | 0/19 | 1/40
Musculoskeletal anomaly (Musculoskeletal and connective tissue disorders) | 1/19 | 0/40
Osteopenia (Musculoskeletal and connective tissue disorders) | 1/19 | 0/40
Apnea (Respiratory, thoracic and mediastinal disorders) | 1/19 | 0/40
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1/19 | 3/40
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0/19 | 1/40
Pulmonary physical finding (Respiratory, thoracic and mediastinal disorders) | 1/19 | 0/40
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1/19 | 2/40
Application site reaction (Skin and subcutaneous tissue disorders) | 0/19 | 1/40
Contact dermatitis (Skin and subcutaneous tissue disorders) | 2/19 | 0/40
Conjunctivitis (Eye disorders) | 1/19 | 0/40
Retinal disorder (Eye disorders) | 1/19 | 1/40
Urinary tract infection (Renal and urinary disorders) | 0/19 | 1/40
Urine abnormality (Renal and urinary disorders) | 1/19 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.